CLINICAL TRIAL: NCT01282580
Title: Omega 3 Fatty Acids and Breast Cancer Prevention: Protective Benefits of Increased Fish Consumption
Brief Title: Dietary Fish and Omega 3 Fatty Acids for Breast Cancer Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-10024; NCI-2012-02933 (Registry Identifier: Clinical Trials Reporting Program)
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: Women at high risk of developing breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary fish (canned salmon, albacore) (Experimental): Fish products: Canned albacore and salmon will be provided at no cost to the patient. Supplies of tuna and salmon will be provided in quantities sufficient for one month of daily intake by the subject. If desired, a subject can request a sufficient amount to allow for preparation of a meal for the family or household at no more than two times per week. Labels or portions of labels from the cans will be collected at the monthly study visits, and canned supplies will be replenished monthly or at more frequent intervals if needed. Subjects will be allowed to keep unused cans.
  Interventions: Other: Dietary fish (canned salmon, albacore)
- Lovaza-Omega 3 fatty acid capsules (Experimental): Lovaza capsules will be provided at no cost to the patient. Pill bottles will be provided to the patient, with the start date and number of pills recorded. The supplement will be provided in sufficient supply for one month at a time. Pill bottles will be collected at monthly follow-up visits, and any unused capsules will be documented and discarded as biohazardous waste.
  Interventions: Dietary Supplement: Lovaza-Omega 3 fatty acid capsules

INTERVENTIONS:
Dietary Supplement: Lovaza-Omega 3 fatty acid capsules — The study will require monthly visits at 0, 1, 2 and 3 months of study intervention. At each visit a fasting serum sample will be obtained, self-report diaries (adverse events, record of omega 3 supplement doses or fish servings taken/missed) will be collected, and pill count / labels from cans of fish will be recorded. Medications and supplements will be reviewed with participants at each monthly visit. At clinic visits at 0 and 3 months, a history and physical examination and breast adipose fine needle aspiration (FNA)will be performed.Omega 3 supplements will be dispensed in monthly amounts.
  Arms: Lovaza-Omega 3 fatty acid capsules
Other: Dietary fish (canned salmon, albacore) — Participants randomized to dietary fish will be asked to incorporate fish in the form of canned albacore and salmon into their diets at four 6 oz servings per week for 3 months. Participants on the dietary fish arm of the study will receive recipes using canned salmon and/or albacore. Sufficient canned salmon/albacore will be available for subjects who wish to prepare a meal for the family/household. Dietary intake will be assessed via 3 day diet records (0 and 3 months) and food frequency questionnaires (0 and 3 months). Verbal and written instructions on how to keep diet records, with food measured or weighed, will be given.
  Other Names: canned fish
  Arms: Dietary fish (canned salmon, albacore)

SUMMARY:
Research studies show that the type of fat in the diet may affect breast cancer risk. Fish oil and fish contain increased amounts of omega 3 fatty acids which appear to stop or slow down the growth and development of breast cancer cells in laboratory studies of mice and breast cancer cells. The use of omega 3 fatty acids to reduce the risk of breast cancer development in humans has not been adequately studied. Eating fish or taking fish oil may increase the amount of omega 3 in the breast, which may lower one's risk of breast cancer development.

Persons in this study with do one of the following: (1) take two capsules daily of omega 3 fatty acid supplements, or (2) eat several servings of canned salmon / tuna per week for a total of three months. Amounts of omega 3 fatty acids in the body's tissues will be measured by blood tests and a small sample of breast fat as obtained by a fine needle aspiration.

This study is supported by funding from the National Fisheries Institute, Food Innovation Center of The Ohio State University, and The Ohio State University Comprehensive Cancer Center.

DETAILED DESCRIPTION:
The primary objectives of this study are to:

i.) Determine the effects of increased fish consumption on serum and breast fat tissue fatty acids in women at high risk for developing breast cancer relative to an omega 3 fatty acid supplement;

ii.) Assess adherence and tolerability of increased dietary intake of fish relative to an omega 3 fatty acid supplement.

Secondary objectives include:

iii.) Evaluate possible correlations between physical factors such as body mass index (BMI) and dietary factors and target tissue effects.

iv.) Explore additional biomarkers as surrogate endpoints to measure effects of fish consumption.

ELIGIBILITY:
Inclusion Criteria:

* Increased risk for breast cancer based on family history, personal history
* Normal mammogram, clinical breast examination in the past 12 months
* >1 year from pregnancy, lactation or chemotherapy

Exclusion Criteria:

* Concurrent malignancy or metastatic malignancy of any kind
* History of a bleeding tendency, use of anticoagulant medications
* Inability to undergo fine needle aspiration of breast adipose tissue
* Chronic use of omega-3 fatty acid supplements or regular consumption of > 2 meals/servings of fish per week within the 3 months prior to entry on the study or any other supplements that might interact with omega-3 fatty acid supplements
* Known sensitivity or allergy to fish
* Standing regimen of full dose aspirin (325 mg/day or more), Non-steroidal anti-inflammatory drugs (NSAIDs) or NSAID-containing products.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Fatty acid profiles of breast adipose tissue | 0 and 3 months

SECONDARY OUTCOMES:
Fatty acid profiles of serum, red blood cell membranes | 0 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa D Yee, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu